CLINICAL TRIAL: NCT02614391
Title: Randomized Controlled Trial to Evaluate Tablet Distraction for Pain Control in Children Underwent Venipuncture
Brief Title: Tablet Distraction for Pain Control During Venipuncture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Principal Investigator, Ronfani Luca, MD, PhD, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 38/12
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Pain Relief
Keywords: Procedural pain; Phlebotomy; Distraction; Videogame; Computer tablet; Child
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active distraction using a tablet (Experimental): Children were admitted in a comfortable room with a parent and started to play with a videogame suitable for their age three minutes before procedure. They continued to play the videogame during venipuncture. The use of a computer tablet permitted to play with one hand only.
  Interventions: Other: Active distraction using a tablet
- Passive distracion (Active Comparator): Children were admitted in a comfortable room with a parent and received various kinds of passive distractions: nurses singing a song, reading a book, blowing bubbles and playing a puppet show. The technique that most engaged the child, was continued during procedure.
  Interventions: Other: Passive distraction

INTERVENTIONS:
Other: Active distraction using a tablet — Playing a videogame using a computer tablet
  Arms: Active distraction using a tablet
Other: Passive distraction — A nurses singing a song, reading a book, blowing bubbles and playing a puppet show
  Arms: Passive distracion

SUMMARY:
Venipuncture is one of the painful procedures most frequently performed in children. Pain and distress management in children, during needle related procedures, is warranted.

The base for pain management starts with behavioural and environmental support and distraction. Distraction is a cognitive strategy trying to divert the child's attention from a noxious stimulus. Active distraction involves the child in a different performance, e.g. playing, during pain procedures. Passive distraction redirects the child's attention to visual or auditory stimuli using toys, songs, movies or blowing bubbles.

Blood-drawing centre is a peculiar setting in which many procedures have to be performed in a limited time. Patients usually arrive without a pharmacological premedication and go away immediately after procedure. In this context distraction is an excellent pain relief tool.

The aim of the study is to compare the effectiveness of an active distraction (playing a videogame using a computer tablet) with a passive distraction technique in pain relief during venipuncture in a blood-drawing centre.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 13 years
* Need for venipuncture
* Informed consent signed by parents or legal guardians

Exclusion Criteria:

* Children with epilepsy
* Use of topical, enteral or parenteral analgesics within 8 hours before the procedure
* Inability to perform venipuncture on hand or arm
* Children with cognitive impairment or unable to report their pain verbally

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pain score recorded by the Faces Pain Scale-Revised (FPS-R) | Intraprocedural (an average of 5 minutes)
  The pain during the procedure will be evaluated using the self-reported FPS-R scale

SECONDARY OUTCOMES:
Success at first attempt | Intraprocedural (an average of 5 minutes)
  Percentage of success at first attempt
Adverse events | Up to 15 minutes after the procedure
  The number and the type of adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Franca Crevatin, RN, Study Chair — IRCCS Burlo Garofolo; Franca Crevatin, RN, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Friuli Venezia Giulia, Italy